CLINICAL TRIAL: NCT04995562
Title: Use of Hyperpolarized 129Xe MR Lung Imaging in Infants
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Xe and Neonates_2019-0810
Record Dates: First submitted 2021-04-12; First posted 2021-08-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Lungs; Developmental Disorder
Keywords: 129 Xe MRI; hyperpolarized xenon; neonates; nasal cannula; HFNC; CPAP; RAM cannula
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: The study includes 2 cohorts: 6 infants on oxygen with nasal cannula, and 6 infants currently requiring respiratory support with high flow nasal cannula (HFNC), continuous positive airway pressure (CPAP) or RAM cannula.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxygen with nasal cannula (Experimental): 6 infants on oxygen with nasal cannula
  Interventions: Drug: 129Xe
- HFNC, CPAP, or RAM cannula (Experimental): 6 infants currently requiring respiratory support with high flow nasal cannula (HFNC), continuous positive airway pressure (CPAP) or RAM cannula
  Interventions: Drug: 129Xe

INTERVENTIONS:
Drug: 129Xe — Inhaled contrast for MRI

SUMMARY:
Abnormalities of the lungs are common in newborns and can include aspiration or infectious pneumonia, respiratory distress syndrome (RDS), bronchopulmonary dysplasia (BPD), pulmonary hypertension (PH), congenital diaphragmatic hernia (CDH), and other abnormalities of lung development. Diagnostic radiography is commonly used in this population to differentiate diagnosis and to assess changes after treatment. While X-ray and CT provide quality imaging, they also expose infants to ionizing radiation. MR imaging offers a safe, non-ionizing alternative. However, imaging lungs via 1H MR is intrinsically difficult due to multiple air-tissue interfaces within the lungs causing local gradients and severe magnetic field susceptibility, which leads to an exceedingly short effective transverse relaxation time (T2*). Additionally, the lungs have low proton density, which along with the short T2* results in low signal to noise ratio, and the physiological motion caused by respiration and cardiac pulsation further reduces lung signal. The development of more powerful hardware, along with faster MRI techniques, has enabled detailed noninvasive 1H MR imaging of pulmonary tissues. Additionally, the development of inhaled hyperpolarized gas MRI has led to breakthroughs in the ability to visualize and quantify regional ventilation and alveolar size.

DETAILED DESCRIPTION:
MRI with hyperpolarized xenon-129 and helium-3 noble gases has been tested and utilized at CCHMC in adults and children over 4 years with a very strong safety record. The safety of both helium-3 and xenon-129 is well known, with 3He being used safely and effectively to image infants, and 129Xe being used extensively in school-age children at CCHMC and elsewhere. Upon inhalation of an anoxic gas mixture, this mixture mixes with the residual volume of standard oxygenated breathing air that remains in the lung even after a normal exhalation, yielding a hypoxic breath. This is performed in the MRI room with pulse oximetry.

The investigators believe, based upon over 2 decades of experience with these noble gases, that the risk of the procedure is very low and primarily relates to the tidal hypoxic inhalation. (The reason for the hypoxic inhalation is because of the depolarizing effects of O2 on the hyperpolarized gas MRI signal.) Thus, an unpublished pilot feasibility study at Cincinnati Children's Hospital was conducted with infants age 0 - 5 months to provide safety data to expand MRI with gases to the neonatal population by pilot testing a brief hypoxic challenge in a controlled setting. The study was conducted in the NICU and included an induced 3-second apnea breath-hold with inhaled nitrogen (N2) while the infant was closely monitored. The study progressed stepwise beginning with 3 infants on room air, 3 infants on oxygen with nasal cannula, then 3 infants currently requiring respiratory support with CPAP or RAM cannula. After each cohort of 3, there was a safety review by the PI and at least one Sub-I who is also a faculty member in the NICU to determine safety before progressing to the next cohort. Results indicate that the procedure was feasible in these populations and was safe. There were no reportable adverse events. Approximately 20 seconds after the breath-hold, there was an expected small transient decline in SpO2 of approximately 5% which quickly (within 5 seconds) returned to baseline, and there were no significant changes in heartrate during the procedure; importantly, no procedure required stopping due to unexpected values. While this pilot study used ultrapure ~100% N2 to induce an apneic period, the degree of apnea will be similar or significantly less with this protocol's xenon apneic periods (Xe concentrations of ~10-100%, and thus will introduce no apneic differences in the proposed study. Safety for this previous pilot study was based upon the much more rigorous clinically accepted hypoxic challenge used to test "fitness-to-fly" done on older infants and children as well as adults. In one research study, the hypoxia challenge test (HCT) was performed on neonates as young as <1 week old with diagnoses of prematurity and BPD. The prospective observational study was carried out on 3 groups of infants: healthy term infants at ≤7 days-old, preterm infants (≥34 weeks CGA) without BPD 2 to 3 days before discharge, and preterm infants with BPD. The infants were placed in a body plethysmograph and inhaled 15% O2 while continuously observed for 20 minutes. If the SpO2 dropped to 85%, the test was stopped and was recorded as a test failure. In Group 1 (full term infants), there was 1 failure out of n=24 (4.2% failure rate). In Group 2 (preterm without BPD), there were 12 failures out of n=62 (19.4% failure rate). In Group 3 (preterm with BPD), there were 16 failures out of n=23 (69.6% failure rate). The BPD infants reached the minimum SpO2 earlier (average 8 minutes) than preterm infants without BPD (average 15 min). While the "fitness-to-fly" test is not routinely performed at Cincinnati Children's, and is typically only utilized at altitude, this previous study with lengthy exposure of the hypoxia challenge is significant in the context of this protocol in that the protocol has significantly less risk (3-second apnea period, as opposed to lengthy hypoxia). Even the BPD cohort had exhibited resilience with an average 8 minute window before desaturation to 85% SpO2.

ELIGIBILITY:
All Cohorts

Inclusion Criteria:

* Male or female
* Any age NICU inpatient who is clinically stable and with adequate temperature control to tolerate MRI as determined by the primary clinical team

Cohort 1

* Age 0 - 6 months
* NICU patient on oxygen with a nasal cannula (≤ 2L per minute) (unchanged - supplemental O2 for minimum 24 hours)
* Maintaining SpO2 > 88% on nasal O2

Cohort 2

* Age 0 - 6 months
* NICU patient who requires a slightly higher level of respiratory support (with High Flow Nasal Cannula > 2L per minute, CPAP, or RAM cannula and O2 unchanged for minimum 24 hours), with FiO2 < 50%.
* Maintaining SpO2 > 88% on nasal O2

Exclusion Criteria:

* General anesthesia within 24 hours prior to MRI or other sedation (e.g. morphine, Versed, fentanyl) within the last 4 hours.
* Extracorporeal membrane oxygenation (ECMO) support
* Evidence of any respiratory infection within 1 week of testing (imaging may be rescheduled for a common viral infection such as a cold).
* Suspected muscular dystrophy or neurologic disorder that may affect lung development.
* Significant genetic or chromosomal abnormalities that may affect lung development
* Congenital heart disease
* Uncontrolled atrial or ventricular arrhythmia
* Open surgical wounds
* Need for inotropic support
* Need for vasodilator agents
* Need for high level of respiratory support (i.e. FiO2 >50%, and/or higher respiratory support than listed in Cohort 2 Inclusion Criteria, such as invasive ventilation).
* Standard MRI exclusion criteria as set forth by the CCHMC Department of Radiology (e.g., contraindicated support/implant equipment that is not MR compatible).
* Infant size not compatible with NICU MRI scanner (~>4.5kg).

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2020-05-06 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation defect percentage (VDP) | 1 day
  To calculate the percentage of the lung that is ventilated with 129Xe gas. This is an indicator of lung ventilation. The lung function outcome will be measured using hyperpolarized 129Xe MRI, wherein hyperpolarized 129Xe is inhaled and its distribution is imaged within the lungs. Different MRI pulse sequences are used to obtain different functional information about the lungs. VDP will be assessed using a 2D spoiled gradient echo sequence.

SECONDARY OUTCOMES:
Apparent diffusion coefficient (ADC) | 1 day
  To calculate the diffusivity coefficient (cm2/s) of the 129Xe gas within the lungs. This is an indicator of regional alveolar microstructure regional distribution in neonatal participants on respiratory support. The lung function outcome will be measured using hyperpolarized 129Xe MRI, wherein hyperpolarized 129Xe is inhaled and its distribution is imaged within the lungs. Different MRI pulse sequences are used to obtain different functional information about the lungs. ADC will be assessed using a 2D diffusion-weighted spoiled gradient echo sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Woods, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Megan Schmitt, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No